CLINICAL TRIAL: NCT01235442
Title: A Randomized Study to Evaluate the Efficacy and Safety of Adding Topical Therapy to Etanercept in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Evaluate Efficacy, and Safety of Topical Therapy and Etanercept in Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20080470
Record Dates: First submitted 2010-10-28; First posted 2010-11-05 (Estimated); Results first posted 2013-10-31 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2015-08

CONDITIONS: Psoriasis
Keywords: Psoriasis; Topical; etanercept; clobetasol propionate
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- etanercept and clobetasol (Experimental): Etanercept 50 mg twice weekly x 12 weeks + clobetasol propionate foam (weeks 11 and 12) then Etanercept 50 mg once weekly x 12 weeks + clobetasol propionate foam (weeks 23 and 24)
  Interventions: Drug: 2=Clobetasol propionate foam
- etanercept (Experimental): Etanercept 50 mg twice weekly x 12 weeks then Etanercept 50 mg once weekly x 12 weeks
  Interventions: Drug: 1=Etanercept

INTERVENTIONS:
Drug: 1=Etanercept — 50 mg SC bi-weekly for 12 weeks followed by 50 mg SC weekly for 12 weeks.
  Arms: etanercept
Drug: 2=Clobetasol propionate foam — 0.05% clobetasol propionate foam applied topically twice daily during two up-to-2 week courses
  Arms: etanercept and clobetasol

SUMMARY:
The primary hypothesis of this trial is that the addition of short courses of clobetasol propionate foam to etanercept monotherapy in subjects with moderate to severe plaque psoriasis will yield greater efficacy compared with etanercept monotherapy, as measured by PASI 75 at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had stable moderate to severe plaque psoriasis for at least 6 months
* Subject has involved BSA ≥ 10% and PASI ≥ 10 at screening and at baseline.
* Subject is a candidate for systemic therapy or phototherapy in the opinion of the investigator

Exclusion Criteria:

* Subject has active guttate, erythrodermic, or pustular psoriasis at the time of the screening visit.
* Subject has evidence of skin conditions at the time of the screening visit (eg, eczema) that would interfere with evaluations of the effect of etanercept and/orclobetasol propionate foam on psoriasis.
* Subject diagnosed with medication-induced or medication exacerbated psoriasis
* Subject has any active Common Toxicity Criteria (CTC) grade 2 or higher infection
* Subject has a significant concurrent medical condition or laboratory abnormalities as defined in the study protocol.
* Subject has used any of the following therapies within 14 days of the first dose: UVB therapy or topical psoriasis therapies other than Class I or II topical steroids.
* Subject has used any of the following therapies within 28 days of the first dose: Class I or II topical steriods, UVA therapy (with or without psoralen), or systemic psoriasis therapies
* Subject has used one or more biologic therapies (other than interleukin (IL)12/IL23 inhibitors) within 3 months of the first dose
* Subject has used an IL-12/IL-23 inhibitor within 6 months of the first dose of etanercept
* Subject has ever used efalizumab (Raptiva®).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Lebwohl MG, Kircik L, Callis Duffin K, Pariser D, Hooper M, Wenkert D, Thompson EH, Yang J, Kricorian G, Koo J. A randomized study to evaluate the efficacy and safety of adding topical therapy to etanercept in patients with moderate to severe plaque psoriasis. J Am Acad Dermatol. 2013 Sep;69(3):385-92. doi: 10.1016/j.jaad.2013.03.031. Epub 2013 May 1. PMID 23643256
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 15 September 2010 through 17 October 2011.
Groups:
- Etanercept Monotherapy: Etanercept 50 mg SC twice weekly for 12 weeks and then 50 mg SC once weekly for 12 weeks (a total of 24 weeks).
- Etanercept + Clobetasol Propionate Foam: Etanercept 50 mg SC twice weekly for 12 weeks and then 50 mg SC once weekly for 12 weeks (a total of 24 weeks). In addition, subjects received topical clobetasol propionate foam twice daily during weeks 11, 12, 23, and 24 as needed until skin was clear of detectable psoriasis (except in proscribed areas).
Period: Overall Study
Arm/Group | Etanercept Monotherapy | Etanercept + Clobetasol Propionate Foam
Started | 297 | 295
Completed | 253 | 251
Not Completed | 44 | 44
Not completed — Lost to Follow-up | 12 | 10
Not completed — Death | 0 | 2
Not completed — Pregnancy | 1 | 1
Not completed — Ineligibility determined | 5 | 4
Not completed — Protocol Violation | 3 | 3
Not completed — Adverse Event | 4 | 6
Not completed — Withdrawal by Subject | 15 | 9
Not completed — Lack of Efficacy | 1 | 3
Not completed — Noncompliance | 1 | 2
Not completed — Administrative decision | 1 | 2
Not completed — Other unspecified | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept Monotherapy | Etanercept + Clobetasol Propionate Foam | Total
Number analyzed (Participants) | 297 | 295 | 592
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.6 (13.7) | 43.7 (14.2) | 44.1 (13.9)
Age, Customized [Number; unit: Participants]
  < 65 years | 273 | 273 | 546
  >=65 years | 24 | 22 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 100 | 201
  Male | 196 | 195 | 391
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 254 | 237 | 491
  Asian | 17 | 19 | 36
  Black or African American | 13 | 18 | 31
  Native Hawaiian or Other Pacific | 0 | 6 | 6
  Mixed Race | 1 | 3 | 4
  American Indian or Alaska Native | 2 | 0 | 2
  Other | 9 | 12 | 21
  Unknown | 1 | 0 | 1
BMI Categorical [Number; unit: Participants]
  ≤ 35 kg/m^2 | 222 | 221 | 443
  > 35 kg/m^2 | 75 | 74 | 149
Psoriasis area severity index (PASI) [Mean (Standard Deviation); unit: Scores on a scale] — PASI is an assessment of psoriasis based on severity of erythema, infiltration, and desquamation as well as area of involvement. The PASI score ranges from 0 to 72. The higher score represents the worse symptom severity.
  Scores on a scale | 18.17 (8.25) | 18.85 (9.16) | 18.51 (8.72)
Psoriasis Body Surface Area(BSA) [Mean (Standard Deviation); unit: %] | 24.09 (17.22) | 25.93 (17.65) | 25.01 (17.44)
Static physician global assessment of psoriasis (sPGA) [Number; unit: Participants] — A physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The sPGA of psoriasis comprises a 6-point scale ranging from 0 (clear) to 5 with increasing severity.
  Participants
    0 | 0 | 0 | 0
    1 | 1 | 1 | 2
    2 | 36 | 46 | 82
    3 | 176 | 164 | 340
    4 | 74 | 74 | 148
    5 | 10 | 8 | 18
    Unknown | 0 | 2 | 2
Patient global assessment of psoriasis [Number; unit: Participants] — A 6-point scale rated by participants ranging from 0 (no symptoms) to 5 (severe symptoms) to indicate his or her symptom severity.
  Participants
    0 | 0 | 0 | 0
    1 | 0 | 3 | 3
    2 | 4 | 6 | 10
    3 | 49 | 58 | 107
    4 | 117 | 95 | 212
    5 | 124 | 127 | 251
    Unkown | 3 | 6 | 9
Dermatology life quality index (DLQI) [Mean (Standard Deviation)] — A skin disease-specific instrument to evaluate health related quality of life ranging from 0 (best possible score) to 30 (worst possible score).
  value | 14.6 (6.9) | 14.1 (7.4) | 14.3 (7.1)
Patient assessment of treatment satisfaction [Number; unit: Participants] — A measure of a participant's level of satisfaction with the medication's control of psoriasis, ranging from "very satisfied" to "very dissatisfied."
  Participants
    Very dissatisfied | 110 | 103 | 213
    Dissatisfied | 40 | 47 | 87
    Neither satisfied nor dissatisfied | 109 | 100 | 209
    Satisfied | 10 | 13 | 23
    Very satisfied | 9 | 11 | 20
    Unknown | 19 | 21 | 40
Psoriatic arthritis [Number; unit: Participants]
  Yes | 84 | 68 | 152
  No | 213 | 227 | 440
Duration of psoriasis [Mean (Standard Deviation); unit: Years] | 17.68 (11.31) | 17.39 (11.89) | 17.53 (11.59)

OUTCOME MEASURES:

1. Primary Outcome: PASI 75 at Week 12
Description: The percentage of participants with the Psoriasis Area and Severity Indexs (PASI) 75 responses at week 12. PASI is an assessment of psoriasis based on severity of erythema, infiltration, and desquamation as well as area of involvement. The PASI score ranges from 0 to 72. The higher score represents the worse symptom severity. A response was considered a 75% reduction in the PASI score from Baseline.
Time Frame: Week 12
Population: Intention-to-Treat with last observation carried forward (LOCF) imputation
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept Monotherapy | Etanercept + Clobetasol Propionate Foam
Number analyzed (Participants) | 297 | 295
Percentage of participants | 48.3 | 65.2
Statistical Analysis 1: Comparison: Etanercept Monotherapy vs Etanercept + Clobetasol Propionate Foam; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Overall significance level for primary and secondary endpoints controlled based on a combination of sequential testing and Hommel procedures; The test is stratified by baseline BMI(=<35 or >35) and prior anti-TNF exposure(Yes or no); Odds Ratio (OR) = 2.05, 95% CI 2-sided [1.46 to 2.87]

2. Secondary Outcome: sPGA (0,1) at Week 12
Description: The percentage of participants achieving sPGA 0 or 1 at week 12. Static physician global assessment of psoriasis (sPGA) is a physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The sPGA of psoriasis comprises a 6-point scale ranging from 0 (clear) to 5 with increasing severity.
Time Frame: Week 12
Population: Intention-to-Treat with last observation carried forward (LOCF) imputation
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept Monotherapy | Etanercept + Clobetasol Propionate Foam
Number analyzed (Participants) | 297 | 295
Percentage of participants | 47.3 | 63.1
Statistical Analysis 1: Comparison: Etanercept Monotherapy vs Etanercept + Clobetasol Propionate Foam; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; The test is stratified by baseline BMI (=<35 or >35) and prior anti-TNF exposure (Yes or No); Odds Ratio (OR) = 1.96, 95% CI 2-sided [1.40 to 2.75]

3. Secondary Outcome: PASI 90 at Week 12
Description: The percentage of participants with the Psoriasis Area and Severity Indexs (PASI) 90 responses at week 12. PASI is an assessment of psoriasis based on severity of erythema, infiltration, and desquamation as well as area of involvement. The PASI score ranges from 0 to 72. The higher score represents the worse symptom severity. A response was considered a 90% reduction in the PASI score from Baseline.
Time Frame: Week 12
Population: Intention-to-Treat with last observation carried forward (LOCF) imputation
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept Monotherapy | Etanercept + Clobetasol Propionate Foam
Number analyzed (Participants) | 297 | 295
Percentage of participants | 19.4 | 29.7
Statistical Analysis 1: Comparison: Etanercept Monotherapy vs Etanercept + Clobetasol Propionate Foam; Test type: Superiority or Other; p = 0.009, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; The test is stratified by baseline BMI (=<35 or >35) and prior anti-TNF exposure (Yes or No); Odds Ratio (OR) = 1.78, 95% CI 2-sided [1.21 to 2.64]

4. Secondary Outcome: Patient Satisfaction at Week 12
Description: Patient assessment of treatment satisfaction status at week 12. It is a measure of a participant's level of satisfaction with the medication's control of psoriasis, ranging from "very satisfied" to "very dissatisfied."
Time Frame: Week 12
Population: PRO analysis set, including all subjects randomized and also complete the baseline and at least 1 of the post-baseline PRO assessment with last observation carried forward (LOCF) imputation
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept Monotherapy | Etanercept + Clobetasol Propionate Foam
Number analyzed (Participants) | 297 | 295
Percentage of participants
  Very dissatisfied | 2.8 | 3.9
  Dissatisfied | 4.9 | 4.3
  Neither satisfied nor dissatisfied | 14.7 | 5.3
  Satisfied | 38.1 | 34.8
  Very satisfied | 39.5 | 51.8
Statistical Analysis 1: Comparison: Etanercept Monotherapy vs Etanercept + Clobetasol Propionate Foam; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; The test is stratified by baseline BMI (=<35 or >35) and prior anti-TNF exposure (Yes or No) with with modified ridit scores

5. Secondary Outcome: Percent PASI Improvement From Baseline at Week 12
Description: The percentage of the improvement in PASI score at week 12 from baseline. PASI is an assessment of psoriasis based on severity of erythema, infiltration, and desquamation as well as area of involvement. The PASI score ranges from 0 to 72. The higher score represents the worse symptom severity.
Time Frame: Week 12
Population: Intention-to-Treat with last observation carried forward (LOCF) imputation
Measure: Mean (Standard Deviation); unit: Percentage of Improvement in PASI score
Arm/Group | Etanercept Monotherapy | Etanercept + Clobetasol Propionate Foam
Number analyzed (Participants) | 297 | 295
Percentage of Improvement in PASI score | 68.18 (29.31) | 76.46 (24.01)
Statistical Analysis 1: Comparison: Etanercept Monotherapy vs Etanercept + Clobetasol Propionate Foam; Test type: Superiority or Other; p < 0.001, van Elteren test — [p-value comment as in outcome 1, analysis 1]; The test is stratified by baseline BMI (=<35 or >35) and prior anti-TNF exposure (Yes or No)

6. Secondary Outcome: PASI 75 at Week 24
Description: The percentage of participants with the Psoriasis Area and Severity Indexs (PASI) 75 responses at week 24. PASI is an assessment of psoriasis based on severity of erythema, infiltration, and desquamation as well as area of involvement. The PASI score ranges from 0 to 72. The higher score represents the worse symptom severity. A response was considered a 75% reduction in the PASI score from Baseline.
Time Frame: Week 24
Population: Intention-to-Treat with last observation carried forward (LOCF) imputation
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept Monotherapy | Etanercept + Clobetasol Propionate Foam
Number analyzed (Participants) | 297 | 295
Percentage of participants | 63.6 | 69.3
Statistical Analysis 1: Comparison: Etanercept Monotherapy vs Etanercept + Clobetasol Propionate Foam; Test type: Superiority or Other; p = 0.135, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; The test is adjusted for baseline BMI (=<35 or >35) and prior anti-TNF (Yes or No); Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.92 to 1.85]

7. Secondary Outcome: sPGA (0,1) at Week 24
Description: The percentage of participants achieving sPGA 0 or 1 at week 24. Static physician global assessment of psoriasis (sPGA) is a physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The sPGA of psoriasis comprises a 6-point scale ranging from 0 (clear) to 5 with increasing severity.
Time Frame: Week 24
Population: Intention-to-Treat with last observation carried forward (LOCF) imputation
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept Monotherapy | Etanercept + Clobetasol Propionate Foam
Number analyzed (Participants) | 297 | 295
Percentage of participants | 54.8 | 61.7
Statistical Analysis 1: Comparison: Etanercept Monotherapy vs Etanercept + Clobetasol Propionate Foam; Test type: Superiority or Other; p = 0.135, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; The test is stratified by baseline BMI (=<35 or >35) and prior anti-TNF exposure (Yes or No); Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.96 to 1.87]

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious adverse events that occurs in 5% participants or more in either arm.
  The numbers of the participants at risk were summarized based on the actual treatment groups, which is different from the randomized treatment groups that were used in the efficacy analysis.
Arm/Group | Etanercept Monotherapy | Etanercept + Clobetasol Propionate Foam
Serious Adverse Events (participants affected / at risk) | 6/301 | 7/288
Other Adverse Events (participants affected / at risk) | 81/301 | 69/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept Monotherapy (N=301) | Etanercept + Clobetasol Propionate Foam (N=288)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Endometritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Tubo-ovarian abscess (Infections and infestations) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept Monotherapy (N=301) | Etanercept + Clobetasol Propionate Foam (N=288)
Nasopharyngitis (Infections and infestations) | 26 | 24
Sinusitis (Infections and infestations) | 14 | 18
Upper respiratory tract infection (Infections and infestations) | 35 | 20
Headache (Nervous system disorders) | 22 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.